CLINICAL TRIAL: NCT04085107
Title: The Moderating Roles of Social Support, Coping Resources and Personality and Mediating Role of Self-esteem on the Impact of Cognitive Deficit on Neuropsychiatric Symptoms Among Persons With Mild Cognitive Impairment: A Mixed-method Sequential Explanatory Design
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Rose Sin Yi Lin, Principal Investigator, Chinese University of Hong Kong
Other Study IDs: 00000
Record Dates: First submitted 2019-09-05; First posted 2019-09-11 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Mild Cognitive Impairment; Behavioral Symptoms
Keywords: mild cognitive impairment; neuropsychiatric symptoms; instrument validation; coping styles; cognitive deficit; neuroticism; social support
MeSH Terms: conditions — Cognitive Dysfunction; Behavioral Symptoms; Cognition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 243 PwMCI
  Interventions: Behavioral: Face-to-face interviews

INTERVENTIONS:
Behavioral: Face-to-face interviews — 243 PwMCI will receive two face-to-face interviews to complete two sets of questionnaires, of which 30 participants will be recruited attend a 1-hour semi-structured interview.

SUMMARY:
This is a sequential mixed study to test the hypothesized models with seven hypotheses of the relationship between cognitive deficit (subject and objective) and neuropsychiatric symptoms (NPS) among persons with mild cognitive impairment (PwMCI). The study will also examine the psychometric properties of the Chinese version of Mild Behavioural Impairment -Checklist (MBI-C).

DETAILED DESCRIPTION:
The primary aim of this study is to test the hypothesized model that explores the moderating roles of neurotic personality, social support and coping style, as well as the mediating role of self-esteem in the relationship between cognitive deficit and NPS. This study will also examine the psychometric properties of the Chinese version of MBI-C.

Specifically, the four objectives of this study are as follows:

1. To examine the relationship between cognitive deficit (subjective and objective) and NPS
2. To examine the moderating roles of the neurotic trait (neuroticism) and coping resources (coping style and social support), as well as the mediating role of self-esteem in the relationship between cognitive deficit and NPS
3. To explore the life experience of PwMCI that help to determine how these factors moderate/ mediate the relationship between cognitive deficit and NPS
4. To examine the psychometric properties of the Chinese version of MBI-C among PwMCI in Hong Kong

This sequential mixed study will be conducted in two non-governmental organization in Hong Kong.

For the first and second objective, a descriptive, cross-sectional, correlational approach will be adopted to test the hypothesized models with seven hypotheses of the relationship between cognitive deficit (subject and objective) and NPS. The moderating roles of personality trait (neuroticism) and coping resources (coping styles and social support), as well as the mediating role of self-esteem in such a relationship, will also be explored.

For the third objective, semi-structured interviews will be adopted to explore the life experience of PwMCI, which help understanding how the proposed factors mediate or moderate the relationship between compromised abilities and NPS.

For the fourth objective, the psychometric properties of the Chinese version of MBI-C will be examined and reported. Internal consistency, 2-week test-retest reliability, factorial validity, concurrent validity and convergent validity will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old or above
* Able to communicate in Cantonese
* Diagnosis with MCI as defined by the following criteria:

  1. Presence of significant cognitive complaints, as defined by more than three complaints on the Memory Inventory for Chinese (MIC), which is a 27-item instrument measuring subjective memory deficit
  2. Abnormal objective cognitive performance defined as < 1.5 standard deviations from age and education matched normal persons on Hong Kong Chinese version of Montreal Cognitive Assessment (HK-MoCA), which is a 12-item instrument measuring cognitive functions
  3. Independence in daily living as evaluated through clinical interview
* Both patients and one of their guardian or family members are consented to participate in the study

Exclusion Criteria:

* With the confirmed diagnosis of any forms of dementia
* With the confirmed diagnosis of psychiatric morbidities, or history with stroke, brain injury and other neurological conditions that may affect cognitive, behavioural and emotional functioning which may confound outcome measurement and limit their participation in the study
* With hearing or visual impairment that may hinder participation in research activities
* Current use of cognitive intervention or electromagnetic stimulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons with mild cognitive impairment in Hong Kong
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2020-03-29 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
Chinese Version of the Neuropsychiatric Inventory Questionnaire (NPI-Q) | Baseline
  NPI-Q is a caregiver-administered instrument that assesses measure the frequency and severity of NPS among the participants.This instrument measures 12 domains including delusion, hallucination, anxiety, depression, euphoria, apathy, disinhibition, irritability and aberrant motor behaviour, sleep disturbance and appetite. The instrument will be completed by an informant to rate the frequency of NPS on a four-point scale (1 - sporadically, 4 - very often) and the severity of NPS on a three-point scale (1 - mild, 3 - severe).
Hong Kong Chinese version of Montreal Cognitive Assessment (HK-MoCA) | Baseline
  This 12-item instrument will be used to measure cognitive functions including visuospatial functions, naming, verbal memory, abstraction, delay memory, calculation and orientation. Total score ranges from 0 to 30, with lower scores indicating more severe cognitive impairment.
Chinese version of Chinese version of Mild Behavioural Impairment -Checklist | Baseline
  This 34-item questionnaire will be used to measure five domains of NPS, including decreased motivation, emotional dysregulation, impulse dyscontrol, social inappropriateness and abnormal perception or thought content. It involves closed-ended questions on the existence of symptoms followed by a 3-point Likert scale on their severity. Total scores of all domains range from 0 to 102, with higher scores indicating more NPS.

SECONDARY OUTCOMES:
Chinese version of Simplified Coping Scale Questionnaire (SCSQ) | Baseline
  This 20-item questionnaire will be adopted to evaluate their attitude towards life events, which could be divided into active (12 items) and passive (eight items) coping styles. Each item is rated at four-point Likert scale, with subscale score are summed from the items in each subscale. A higher subscale score indicates more frequent use of the coping style.
Chinese version of Multidimensional Scale of Perceived Social Support (MSPSS-C) | Baseline
  This 12-item instrument measures the availability of support from family (4 items) and friends (8 items) on a seven-point Likert scale with total scores range from 12 to 48. Higher scores indicate a higher level of perceived social support.
Chinese version of the neuroticism subscale of NEO Personality Inventory (NEO-PI) | Baseline
  This 12-item neuroticism subscale will be adopted to measure neuroticism over manageability, comprehensibility and meaningfulness on a five-point Likert scale. Total scores range from 0 to 48, with higher scores indicating a more neurotic personality.
Rosenberg self-esteem scale (RSES) | Baseline
  The 10-item scale will be adopted to evaluate the sense of self-worth through five positive and five negative statements on a four-point Likert scale, all items are summed to total scores that range from 10 to 40, with a higher score indicating higher level of self-esteem.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong